CLINICAL TRIAL: NCT02566941
Title: Neuromuscular Electrical Stimulation in the Critically Ill
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of human ressources
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Jacques DEVRIENDT, Head of clinic, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CHUB-SNM001
Record Dates: First submitted 2015-08-14; First posted 2015-10-02 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Polyneuropathy
Keywords: critical illness polyneuropathy; critical illness myopathy; neuromuscular electrical stimulation; intensive care unit acquired weakness; prevention of critical illness polyneuropathy
MeSH Terms: conditions — Polyneuropathies

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stimulated (Experimental): Patients included in the 'stimulated' group will be stimulated at the level of the quadriceps twice a day, bilaterally and simultaneously, five days per week from Monday to Friday (Stimulator: Gymna Belgium, DUO 400). The stimulation protocol (rectified alternating current; frequency, 75 Hz; intensity, 0-80 mA; pulse duration, 350 microseconds) is the one proposed by the manufacturer for atrophy prevention. The intensity of the electrical current will be gradually increased, without exceeding 80mA or the pain threshold of the patient.
  Interventions: Device: Gymna Belgium, DUO 400 (Neuromuscular electrical stimulation)
- Control (No Intervention)

INTERVENTIONS:
Device: Gymna Belgium, DUO 400 (Neuromuscular electrical stimulation)
  Arms: Stimulated

SUMMARY:
Neuromuscular stimulation (NMES) has been used for several years in the rehabilitation of COPD (chronic obstructive pulmonary disease) patients (among others) to improve their resistance to efforts in everyday life. In patients in intensive care, it seems to improve strength, reduce the loss of muscle mass, prevent the development of CIP / CIM (Critical illness polyneuropathy / critical illness myopathy) and perhaps even reduce ventilation days, with expected effects on the duration of hospitalization and the long-term functional outcome. Although its use could sometimes be limited by the development of peripheral edema and use of vasoconstrictors, the main advantage of this technique is the possibility of being used very early, even in patients that require deep sedation . This is extremely important given that the muscular atrophy process already starts 18h after the onset of invasive ventilation and as signs of impaired nerve transmission are developed in one third of patients at risk within 72 hours.

The purpose of the study is to assess the effects, in the short and medium term, of early neuromuscular stimulation in patients who are at higher risk of developing a critical illness polyneuropathy (CIP) / critical illness myopathy (CIM) spectrum disease.

This is a randomized controlled single-blind study comparing a group of patients submitted to NMES early (up to 5 days after admission) versus a control group unstimulated.

ELIGIBILITY:
Inclusion Criteria:

* Admission in the ICU of the Brugmann Hospital (Unit 1020) with an intended ICU stay superior to 3 days
* Aged over 18 years
* Respiratory assistance needed (invasive and non-invasive ventilation, CPAP or Optiflow and PaO2(arterial oxygen pressure)/FiO2(fraction of inhaled oxygen)<200mmHg)
* SAPSII (Simplified Acute Physiology Score) between entre 35 et 70.

Exclusion Criteria:

Definitive exclusion criteria:

* patients bearing a pacemaker or an AICD (automatic implantable cardioverter/defibrillator )
* BMI superior to 35
* serious neuromuscular pathologies or alterations in the inferior members that make both tights stimulation impossible
* pregnant women
* patients admitted from Friday evening to Sunday morning

Temporary exclusion criteria:

* Hemodynamic instability (even with filling up and amines: noradrenaline > 0.5y/kg/min and/or dobutamine >5y/kg/min and/or adrenaline ivc)
* Extreme severity with suspicion of death within the first 24 h
* PIC > 20 cmH2O
* Severe agitation (RASS > +1)
* Curare utilisation within the last 24h

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Duration of respiratory support | Patients will be followed for the duration of their intensive care unit stay.The average duration of an intensive care unit stay in the CHU Brugamnn Hospital in 2014, all pathologies mixed, is 6 days.
  The duration of ventilatory support is defined as the time in days, during which the patient requires invasive media type (continuous or not, intubation or tracheotomy and need the help of the respirator) or noninvasive (discontinuous or CPAP NIV (continuous positive airway pressure, noninvasive ventilation)- dependence). This will be assessed during the entire length of stay of the patient inside the intensive care unit (ICU).
Length of stay in the intensive care unit | Patients will be followed for the duration of their intensive care unit stay.The average duration of an intensive care unit stay in the CHU Brugamnn Hospital in 2014, all pathologies mixed, is 6 days.
  Measured in days
Type of hospital discharge | At hospital discharge, within a maximum of two years (approximate study length).
  Back to home or to a specialized long term care structure

SECONDARY OUTCOMES:
cross-sectional area of the rectus femoris | First day in ICU
  The quadriceps muscle mass will be assessed using an ultrasound system (PHILIPS, VIVIDS5).
cross-sectional area of the rectus femoris | Third day in ICU
  The quadriceps muscle mass will be assessed using an ultrasound system (PHILIPS, VIVIDS5).
cross-sectional area of the rectus femoris | Fifth day in ICU
  The quadriceps muscle mass will be assessed using an ultrasound system (PHILIPS, VIVIDS5).
cross-sectional area of the rectus femoris | Seventh day in ICU
  The quadriceps muscle mass will be assessed using an ultrasound system (PHILIPS, VIVIDS5).
cross-sectional area of the rectus femoris | The day the patient is discharged from the intensive care unit. The average duration of an intensive care unit stay in the CHU Brugamnn Hospital in 2014, all pathologies mixed, is 6 days.
  The quadriceps muscle mass will be assessed using an ultrasound system (PHILIPS, VIVIDS5).
Force index - Grip test | Patients will be followed for the duration of their intensive care unit stay.The average duration of an intensive care unit stay in the CHU Brugamnn Hospital in 2014, all pathologies mixed, is 6 days.
  The "Grip Test" involves measuring the grip force developed by the hand of the patient, using a dynamometer (Neugen Medicals MODEL EH 101). This test will be conducted as soon as possible aka when the patient has -1 ≤ RASS ≤ 1, is sufficiently collaborating and little sedated.
Force index - Grip test | The day the patient is discharged from the intensive care unit. The average duration of an intensive care unit stay in the CHU Brugamnn Hospital in 2014, all pathologies mixed, is 6 days.
  The "Grip Test" involves measuring the grip force developed by the hand of the patient, using a dynamometer (Neugen Medicals MODEL EH 101). This test will be performed on the day the patient is discharged from the intensive care unit.
Force index - Bike | Patients will be followed for the duration of their intensive care unit stay.The average duration of an intensive care unit stay in the CHU Brugamnn Hospital in 2014, all pathologies mixed, is 6 days.
  The bike (Neugen Medicals MODEL EH 101) is a true "bike room" which facilitates active and passive mobilization of bedridden patients and allows, among other things, to measure the force developed by the patients and the ratio between active and passive labor work.This test will be conducted as soon as possible aka when the patient has -1 ≤ RASS ≤ 1, is sufficiently collaborating and little sedated.
Force index - Bike | The day the patient is discharged from the intensive care unit. The average duration of an intensive care unit stay in the CHU Brugamnn Hospital in 2014, all pathologies mixed, is 6 days.
  The bike (Neugen Medicals MODEL EH 101) is a true "bike room" which facilitates active and passive mobilization of bedridden patients and allows, among other things, to measure the force developed by the patients and the ratio between active and passive labor work.This will be measured at patient discharge from ICU
Electromyogram | First day of ICU admission
  The Electrical conduction of nerves fibula will be assessed to detect nerve damage. A positive test will involve a complete electrophysiological monitoring by a specialist.
Electromyogram | Third day of ICU admission
  The Electrical conduction of nerves fibula will be assessed to detect nerve damage. A positive test will involve a complete electrophysiological monitoring by a specialist.
Electromyogram | Fifth day of ICU admission
  The Electrical conduction of nerves fibula will be assessed to detect nerve damage. A positive test will involve a complete electrophysiological monitoring by a specialist.
Electromyogram | Seventh day of ICU admission
  The Electrical conduction of nerves fibula will be assessed to detect nerve damage. A positive test will involve a complete electrophysiological monitoring by a specialist.
Electromyogram | The day the patient is discharged from the intensive care unit. The average duration of an intensive care unit stay in the CHU Brugamnn Hospital in 2014, all pathologies mixed, is 6 days.
  The Electrical conduction of nerves fibula will be assessed to detect nerve damage. A positive test will involve a complete electrophysiological monitoring by a specialist.
Physical Function ICU Test score (PFIT-s) | Patients will be followed for the duration of their intensive care unit stay.The average duration of an intensive care unit stay in the CHU Brugamnn Hospital in 2014, all pathologies mixed, is 6 days.
  This simple functional test was developed to measure the functional abilities of patients severely debilitated that are found in the ICU. It consists in assessing four different levels of physical ability: the bending force of the shoulder and knee extension in sitting position, measured with the Oxford scale; the level of assistance needed to move from a sitting position to a standing position; and the ability to stand and walk on site. Patients will be tested as soon as possible aka when the patient has: -1 ≤ RASS ≤ 1, is sufficiently collaborating and not heavily sedated.
Physical Function ICU Test score (PFIT-s) | the day the patient is discharged from the intensive care unit. The average duration of an intensive care unit stay in the CHU Brugamnn Hospital in 2014, all pathologies mixed, is 6 days.
  This simple functional test was developed to measure the functional abilities of patients severely debilitated that are found in the ICU. It consists in assessing four different levels of physical ability: the bending force of the shoulder and knee extension in sitting position, measured with the Oxford scale; the level of assistance needed to move from a sitting position to a standing position; and the ability to stand and walk on site.
Six minutes Walking Test | the day the patient is discharged from the hospital, within a maximum of 2 years (approximate total study length)
  The 6-minute walk test is a validated and commonly used test to assess submaximal functional capacity; the test is conducted according to the guidelines of the American Thoracic Society.
Six minutes Walking Test | one year after the day of admission to the intensive care unit
  The 6-minute walk test is a validated and commonly used test to assess submaximal functional capacity; the test is conducted according to the guidelines of the American Thoracic Society.
MOS SF-36 | the day the patient is discharged from the hospital, within a maximum of two years (approximated study lenght)
  The MOS SF-36 questionnaire will be proposed to patients on the day of hospital discharge and one year after the day of admission to the ICU, to assess their quality of life.
MOS SF-36 | one year after the day of admission to the intensive care unit
  The MOS SF-36 questionnaire will be proposed to patients on the day of hospital discharge and one year after the day of admission to the ICU, to assess their quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Devriendt, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

REFERENCES:
- [Background] Dal-Pizzol F, Ritter C. Functional disability 5 years after ARDS. N Engl J Med. 2011 Jul 21;365(3):274-5; author reply 275-6. doi: 10.1056/NEJMc1105509. No abstract available. PMID 21774725
- [Background] Batt J, dos Santos CC, Cameron JI, Herridge MS. Intensive care unit-acquired weakness: clinical phenotypes and molecular mechanisms. Am J Respir Crit Care Med. 2013 Feb 1;187(3):238-46. doi: 10.1164/rccm.201205-0954SO. Epub 2012 Nov 29. PMID 23204256
- [Background] Hermans G, De Jonghe B, Bruyninckx F, Van den Berghe G. Interventions for preventing critical illness polyneuropathy and critical illness myopathy. Cochrane Database Syst Rev. 2014 Jan 30;2014(1):CD006832. doi: 10.1002/14651858.CD006832.pub3. PMID 24477672
- [Background] Maddocks M, Gao W, Higginson IJ, Wilcock A. Neuromuscular electrical stimulation for muscle weakness in adults with advanced disease. Cochrane Database Syst Rev. 2013 Jan 31;(1):CD009419. doi: 10.1002/14651858.CD009419.pub2. PMID 23440837
- [Background] Dirks ML, Wall BT, Snijders T, Ottenbros CL, Verdijk LB, van Loon LJ. Neuromuscular electrical stimulation prevents muscle disuse atrophy during leg immobilization in humans. Acta Physiol (Oxf). 2014 Mar;210(3):628-41. doi: 10.1111/apha.12200. Epub 2013 Dec 12. PMID 24251881
- [Background] Routsi C, Gerovasili V, Vasileiadis I, Karatzanos E, Pitsolis T, Tripodaki E, Markaki V, Zervakis D, Nanas S. Electrical muscle stimulation prevents critical illness polyneuromyopathy: a randomized parallel intervention trial. Crit Care. 2010;14(2):R74. doi: 10.1186/cc8987. Epub 2010 Apr 28. PMID 20426834
- [Background] Burke D, Gorman E, Stokes D, Lennon O. An evaluation of neuromuscular electrical stimulation in critical care using the ICF framework: a systematic review and meta-analysis. Clin Respir J. 2016 Jul;10(4):407-20. doi: 10.1111/crj.12234. Epub 2014 Nov 26. PMID 25353646
- [Background] Hirose T, Shiozaki T, Shimizu K, Mouri T, Noguchi K, Ohnishi M, Shimazu T. The effect of electrical muscle stimulation on the prevention of disuse muscle atrophy in patients with consciousness disturbance in the intensive care unit. J Crit Care. 2013 Aug;28(4):536.e1-7. doi: 10.1016/j.jcrc.2013.02.010. Epub 2013 Apr 3. PMID 23561945
- [Background] Segers J, Hermans G, Bruyninckx F, Meyfroidt G, Langer D, Gosselink R. Feasibility of neuromuscular electrical stimulation in critically ill patients. J Crit Care. 2014 Dec;29(6):1082-8. doi: 10.1016/j.jcrc.2014.06.024. Epub 2014 Jun 30. PMID 25108833
- [Background] Levine S, Nguyen T, Taylor N, Friscia ME, Budak MT, Rothenberg P, Zhu J, Sachdeva R, Sonnad S, Kaiser LR, Rubinstein NA, Powers SK, Shrager JB. Rapid disuse atrophy of diaphragm fibers in mechanically ventilated humans. N Engl J Med. 2008 Mar 27;358(13):1327-35. doi: 10.1056/NEJMoa070447. PMID 18367735
- [Background] Latronico N, Bertolini G, Guarneri B, Botteri M, Peli E, Andreoletti S, Bera P, Luciani D, Nardella A, Vittorielli E, Simini B, Candiani A. Simplified electrophysiological evaluation of peripheral nerves in critically ill patients: the Italian multi-centre CRIMYNE study. Crit Care. 2007;11(1):R11. doi: 10.1186/cc5671. PMID 17254336
- [Background] Seymour JM, Ward K, Sidhu PS, Puthucheary Z, Steier J, Jolley CJ, Rafferty G, Polkey MI, Moxham J. Ultrasound measurement of rectus femoris cross-sectional area and the relationship with quadriceps strength in COPD. Thorax. 2009 May;64(5):418-23. doi: 10.1136/thx.2008.103986. Epub 2009 Jan 21. PMID 19158125
- [Background] Latronico N, Nattino G, Guarneri B, Fagoni N, Amantini A, Bertolini G; GiVITI Study Investigators. Validation of the peroneal nerve test to diagnose critical illness polyneuropathy and myopathy in the intensive care unit: the multicentre Italian CRIMYNE-2 diagnostic accuracy study. F1000Res. 2014 Jun 11;3:127. doi: 10.12688/f1000research.3933.3. eCollection 2014. PMID 25309729
- [Background] Skinner EH, Berney S, Warrillow S, Denehy L. Development of a physical function outcome measure (PFIT) and a pilot exercise training protocol for use in intensive care. Crit Care Resusc. 2009 Jun;11(2):110-5. PMID 19485874
- [Background] Denehy L, de Morton NA, Skinner EH, Edbrooke L, Haines K, Warrillow S, Berney S. A physical function test for use in the intensive care unit: validity, responsiveness, and predictive utility of the physical function ICU test (scored). Phys Ther. 2013 Dec;93(12):1636-45. doi: 10.2522/ptj.20120310. Epub 2013 Jul 25. PMID 23886842
- [Background] Parry SM, Denehy L, Beach LJ, Berney S, Williamson HC, Granger CL. Functional outcomes in ICU - what should we be using? - an observational study. Crit Care. 2015 Mar 29;19(1):127. doi: 10.1186/s13054-015-0829-5. PMID 25888469